CLINICAL TRIAL: NCT02337582
Title: Pilot Study for Implementing Breast Cancer Early Detection Programs in Colombia
Brief Title: Colombian Screening Mammography Project
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fred Hutchinson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Screening
Other Study IDs: SAC110001; 6465 (Other: FHCRC)
Record Dates: First submitted 2015-01-09; First posted 2015-01-13 (Estimated); Last update posted 2015-01-13 (Estimated); Status verified 2015-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Intervention (Active Comparator)
  Interventions: Other: Opportunistic Breast cancer screening
- Control (Other)
  Interventions: Other: Usual Care

INTERVENTIONS:
Other: Opportunistic Breast cancer screening — Opportunistic breast screening offered to women attending clinics for non-breast health issues
  Arms: Intervention
Other: Usual Care — No breast screening was explicitly offered to women attending clinics for non-breast health issues, unless the health care provider felt that it was appropriate
  Arms: Control

SUMMARY:
A cluster randomized controlled trial was performed in Bogotá, Colombia between 2007-2008 to evaluate the effects of an opportunistic (hospital-based) screening program (intervention) vs. usual care (control) in which 26 clinics were randomized to an intervention (N=13) or control arm (N=13). At intervention clinics general practitioners were instructed to perform clinical breast examination (CBE) on all women aged 50-69 years attending clinics for non-breast health related issues, and to refer them for mammographic screening. Physicians from control clinics were not specifically instructed to perform breast-screening or refer women for mammography, but could do so if they thought it appropriate ('usual care'). Women were followed for 2 years post-randomization.

ELIGIBILITY:
Inclusion Criteria:

Female Aged 50-69 Resident in Bogotá, Colombia or surrounding cities; Had not had a mammogram in the previous two years; No history of breast cancer Attending health-centers for reasons unrelated to breast health

Exclusion Criteria:

* see above

Ages: 50 Years to 69 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 15855 (Actual)
Dates: Start 2007-01; Primary Completion 2012-12 (Actual); Study Completion 2014-08 (Actual)

PRIMARY OUTCOMES:
Breast cancer Incidence | Two years
  Comparing incidence of breast cancer in women randomized to the opportunistic breast screening arm, compared to women in the control arm.

CONTACTS AND LOCATIONS:
Locations (1):
- Fred Hutchinson Cancer Research Center, Seattle, Washington, United States

REFERENCES:
- [Derived] Murillo R, Diaz S, Perry F, Poveda C, Pineros M, Sanchez O, Buitrago L, Gamboa O, Lozano T, Yu H, Wang CY, Duggan C, Thomas DB, Anderson BO. Increased breast cancer screening and downstaging in Colombian women: A randomized trial of opportunistic breast-screening. Int J Cancer. 2016 Feb 1;138(3):705-13. doi: 10.1002/ijc.29801. Epub 2015 Sep 2. PMID 26264446